CLINICAL TRIAL: NCT05898568
Title: Virtual Reality in Hand Peripheral Nerve Injuries Effectiveness of Based Movement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Serkan Kablanoğlu, occupational therapist, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-66175679-514.13.02-960185
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Peripheral Nerve Injury, Virtual Reality, Rehabilitation
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental: virtual reality (Experimental): In addition to routine hand care programs for 4 weeks, 5 days, 40 minutes a day, 20 sessions (4 weeks, 5 days, 20 minutes) virtual reality based movement therapy program will be applied.
  Interventions: Device: virtual reality
- control:routine treatment (Active Comparator): 20 sessions (4 weeks, 5 days a week, 60 minutes) routine hand rehabilitation program will be implemented.
  Interventions: Behavioral: routine treatment

INTERVENTIONS:
Device: virtual reality — In addition to the routine hand rehabilitation programs for 4 weeks, 5 days, 40 minutes a day, 20 sessions (4 weeks, 5 days a week, 20 minutes) virtual reality based movement therapy program will be applied.
  Arms: experimental: virtual reality
Behavioral: routine treatment — 20 sessions (4 weeks, 5 days a week, 60 minutes) routine hand rehabilitation program will be applied.
  Arms: control:routine treatment

SUMMARY:
The aim of this study is to investigate the effectiveness of virtual reality-based motion therapy in peripheral nerve injuries in the hand.

ELIGIBILITY:
Inclusion Criteria:

* ıt was operated in the early period with the diagnosis of peripheral nerve injury in the postoperative hand.
* clinical impression was made.
* out patient with median, ulnar, and radial nerve repair.
* completed the 6th postoperative week.

Exclusion Criteria:

* Those who have communication problems and users
* With the musculoskeletal system, the additional passage, rheumatological, etc., where they are located.

those with the disease

- Patients with multiple traumas

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Jebsen Taylor Hand Function Test | from baseline to the end of the treatment (4 week)
  Used to assess upper extremity functions. Activities are evaluated on a time basis.
visual analog scale (VAS) | from baseline to the end of the treatment (4 week)
  marks the severity of pain between 0 and 10.
duruöz hand index | from baseline to the end of the treatment (4 week)
  kitchen work, evaluates cleaning, workplace and other activities of daily living. The total score is between 0-90.
Sammes Weinstein Monofilament Test (SWMT) | from baseline to the end of the treatment (4 week)
  sensory threshold is used for assessment.sensed monofilament values will be collected and recorded. The highest total score will be considered as 15.
Questionnaire Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) | from baseline to the end of the treatment (4 week)
  activity participation level will be assessed by Q-DASH.Each question will be scored between 1-5 points (1: no difficulty, 2: mild difficulty, 3: medium difficulty, 4: extreme difficulty, 5: not at all). The total score will be recorded.
Jamar dynamometer | from baseline to the end of the treatment (4 week)
  Jamar dynamometer will be used for grip strength. 3 repetitive measurements will be made and the average will be recorded.(in kilograms)

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli University, Kocaeli, Arızlı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No